CLINICAL TRIAL: NCT03352479
Title: Keeping Your Children and Home Safe Through Return and Disposal of Unused Opioids
Brief Title: Safe Return and Disposal of Unused Opioids
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: this is an observational project and doesn't not meet any of the four criteria required for listing on clinical trials.gov
Sponsor: Baylor College of Medicine (Other)
Collaborators: Chandrakantan (Unknown)
Responsible Party: Principal Investigator, Adam Adler MD, MS, FAAP, Assistant Professor of Anesthesiology, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H42451
Record Dates: First submitted 2017-11-21; First posted 2017-11-24 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Opioid Use; Opioid Dependence; Opioid Abuse, Unspecified
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Each participant will be given on envelope to return unused opioids
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Opioids Prescribed (Other): Each participant in the study will be given an envelope for return of unused opioids. The percentage of returned number of opioids will be calculated based on the number prescribed
  Interventions: Other: Opioid Return

INTERVENTIONS:
Other: Opioid Return — Calculate the percentage of prescribed to returned opioids

SUMMARY:
The opioid epidemic in the United States has become a clear health and safety concern for our children and families. Opioids given to our patients for the treatment of pain that go unused after the immediate post operative period pose a major hazard when left in the home unattended. Opioids can be accidentally ingested by small children or deliberately ingested by pre-teens and adolescents leading to major morbidity and or death. Additionally, studies have shown that many people addicted to opioids/narcotics have become so due to ingestion of medically prescribed drugs. Finally, there has been an increase number of home robberies specifically with the intent to steal prescription drugs. Removal of unused medication from the home is an important public safety concern to protect our patients, families and friends. The Sharps Co (R), offers a product called Takeaway Medication Recovery System. This product allows individuals to put unused opioids in a pre-paid envelope which is returned to the company through the postal system and properly incinerated. This provides safe disposal in accordance with the Environmental Protection Agency (EPA) to protect the water table from contamination by drugs disposed of my other means. This system through the Sharps Co would allow for de-identified tracking of returned drugs.

DETAILED DESCRIPTION:
Participants identified by the PI and participating research staff/coordinators that will receive opioids following discharge will be approached. The participant information sheet will be provided to the parents/legal guardian and explained. The consenting study coordinator will review the potential risks of opioids as described in the information sheet. A brief demonstration of the TakeAway envelope will be provided. The participants will be instructed that there is absolutely no cost to them or their family and that the envelope is pre-paid and that all returned or unreturned contents are strictly confidential. A few brief demographic questions will be asked and are completely optional. The participant will be asked for an email and contacted 15 days and 30 days following the procedure. The email will strictly be a reminder to return all un-used medication using the provided envelope Or an optional response reporting nothing to return. If participants do not have an email or do not wish to be contacted, they may still enroll in the study. The entire peri-operative period will progress in the usual manner.

Each envelope has a serial number that will be recorded during enrollment - the company provides access to ascertain exactly how many pills are returned. This access is strictly provided to the PI. The company will have no patient information and therefore only the PI will be able to track the serial number to the patient. The PI and research staff will record the number of pills prescribed to the patient to allow the research team to calculate the percentage of pills returned.

ELIGIBILITY:
Inclusion Criteria:

* All patients being prescribed opioids at discharge in the Clinical Care Center/Wallace Tower Surgical Center or at the Woodlands Campus who have undergone a surgical procedure.

Exclusion Criteria:

* Parental Refusal to participate Patients not being prescribed opioids for discharge Patients on chronic opioid therapy/chronic pain patients International patients returning abroad (these takeaway envelopes are only paid through the 50 US states, DC and Puerto Rico)

Max Age: 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-07-30 (Estimated)

PRIMARY OUTCOMES:
% of prescribed unused opioids returned | six months
  Calculate the percentage of opioids that are prescribed that are safely returned by participants and their families

REFERENCES:
- [Derived] Adler AC, Yamani AN, Sutton CD, Guffey DM, Chandrakantan A. Mail-Back Envelopes for Retrieval of Opioids After Pediatric Surgery. Pediatrics. 2020 Mar;145(3):e20192449. doi: 10.1542/peds.2019-2449. Epub 2020 Feb 12. PMID 32051219